CLINICAL TRIAL: NCT02269761
Title: Prospective Evaluation With Ultrasound of Emergency Department Patients Presenting With Cough or Dyspnea
Brief Title: Chest Ultrasound of ER Patients With Cough or SOB
Status: Terminated | Type: Observational
Why Stopped: The patients were too sick to consent and we couldn't recruit enough to continue the study
Sponsor: University of Washington (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Theodore Dubinsky, Professor, Radiology, University of Washington
Other Study IDs: 47935
Record Dates: First submitted 2014-10-03; First posted 2014-10-21 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cough; Dyspnea; Wheezing
Keywords: Emergency Departments; Chest; Lung; Cough; Dyspnea; Wheezing; Ultrasound; Ultrasonography
MeSH Terms: conditions — Cough; Dyspnea; Respiratory Sounds; Emergencies | interventions — Transducers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Nuvis Diagnostic Ultrasound System — Ultrasound of the chest
  Other Names: Diagnostic ultrasound system and transducers; C5-2 curve linear array USB transducer

SUMMARY:
Acute dyspnea (shortness of breath) is a common complaint for patients presenting to the Emergency Department (ED). The chest radiograph (CXR) has been the mainstay in evaluating patients with shortness of breath and often provides the timely diagnosis of pneumonia, pneumothorax, pulmonary edema, among other primary diseases of the lung. There are limitations with chest radiograph such as large body mass (e.g, obesity) and patient positioning. On occasion, chest radiography findings are difficult to interpret. Lung ultrasonography may offer a means of clarifying ambiguous results.

The objective of this study to determine the usefulness of point of care lung ultrasound in evaluating patients presenting to the ED with shortness of breath, cough and/or wheezing.

DETAILED DESCRIPTION:
Acute dyspnea (shortness of breath) is a common complaint for patients presenting to the Emergency Department (ED). The chest radiograph (CXR) has been the mainstay in evaluating patients with shortness of breath and often provides the timely diagnosis of pneumonia, pneumothorax, pulmonary edema, among other primary diseases of the lung. There are limitations with chest radiograph such as large body mass (e.g, obesity) and patient positioning. On occasion, chest radiography findings are difficult to interpret. Lung ultrasonography may offer a means of clarifying ambiguous results. Advantages of ultrasound include real-time immediate evaluation, it is non-invasive and does not use radiation.

The investigators seek to perform a prospective evaluation of patients presenting to the University of Washington Medical Center ED for cough, wheezing and/or shortness of breath.

The objective of this study to determine the usefulness of point of care lung ultrasound in evaluating patients presenting to the ED with shortness of breath, cough and/or wheezing.

The specific aim of this study is to further define the utility of point-of-care ultrasound in the evaluation of emergency department patients presenting with cough, wheezing and/or shortness of breath. The investigators will compare ultrasound results to radiograph and tomography results when available, and to the physicians initial impression.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the Emergency Department with cough, wheezing and/or dyspnea (shortness of breath)
* Referred for CXR and/or CT scan

Exclusion Criteria:

* Life threatening medical condition requiring immediate treatment
* Unable to sit up for a chest ultrasound
* Unable to consent
* Pregnant
* Unable to speak, read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department (ED) patients with shortness of breath (SOB)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
B-lines on chest ultrasound as a predictor of pulmonary edema and/or pneumonia | Up to 1 week
  Results from the study ultrasound will be correlated with other imaging results and the emergency physicians initial impression.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore J Dubinsky, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States